CLINICAL TRIAL: NCT04953754
Title: Melatonin and Vaccine Response, Immunity, and Chronobiology Study (MAVRICS): The Impact of Sleep, Circadian Health, and Melatonin on Vaccine Immunogenicity and Outcomes
Brief Title: Melatonin and Vaccine Response, Immunity, and Chronobiology Study
Acronym: MAVRICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rachel Lee, Service Chief, Allergy, Immunology & Immunizations, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMRC.2021.0006
Record Dates: First submitted 2021-06-04; First posted 2021-07-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Vaccine Response; Sleep; Circadian Rhythm Disorders
Keywords: Sleep; Circadian health; Vaccine immunogenicity; Melatonin
MeSH Terms: conditions — Chronobiology Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Prospective open label melatonin compared to control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Melatonin Group (Experimental): This group will get melatonin 5mg nightly
  Interventions: Dietary Supplement: Melatonin; Device: Phillips Actiwatch Spectrum Plus
- Control Group (Active Comparator): This group will not get any treatment (melatonin)
  Interventions: Device: Phillips Actiwatch Spectrum Plus

INTERVENTIONS:
Dietary Supplement: Melatonin — The melatonin group will receive 5mg melatonin nightly
  Arms: Melatonin Group
Device: Phillips Actiwatch Spectrum Plus — Both groups will be monitored by the FDA-cleared Actigraph

SUMMARY:
This study will evaluate the impact of sleep, circadian health and melatonin on flu vaccine immunogenicity.

DETAILED DESCRIPTION:
Vaccination is critical to public health and disease prevention. However, despite the many scientific advancements and vaccines on the market, they are not always fully effective. Adjuvants are often used to boost immunity, but they are associated with more side effects, possible allergic reactions and public mistrust that supports vaccine hesitancy. Many factors affect vaccine efficacy and host immunity. Sleep, circadian health and melatonin have been studied in the past to affect immune response to vaccines and infection. Patient education about better sleep habits and/or melatonin use are potentially safe, cost effective, and accessible interventions that may improve host immunity and vaccine effectiveness. However, neither have been studied rigorously and at this time, are not actively implemented in the clinical arena. Hence, we propose a study comparing vaccine immunogenicity based on sleep quality, chronotype, and exogenous melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Eligible to receive flu vaccination (at military hospital, DEERS eligible)

Exclusion Criteria:

* Allergy or contraindication to getting flu vaccine
* Pregnancy or likelihood of getting pregnant in next few weeks
* Medical history of doctor diagnosed immune-compromising condition (HIV/AIDS, cancer, diabetes, significant cardiovascular disease) or doctor diagnosed sleep disorder (insomnia, narcolepsy).*Sleep apnea is an exclusion unless stable on treatment with cpap or oral device for more than3 months.
* Currently taking any immune suppressants or immunomodulating treatments (systemic corticosteroids, chemotherapy, etc, within the past 3 months) or sleep medication or supplement (including over the counter medications and melatonin, within the past 1 month).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Anti-influenza antibody titers | 14-21 days post vaccination
  Seroconversion and titer >=1:40 post-vaccination
Cell-mediated immunity | 14-21 days post vaccination
  ELISpot (secretion of Interferon-gamma and Granzyme B with restimulation by influenza viral antigens), Flow cytometry to determine CD4+ and CD8+ T cell producing IFN(g) with influenza viral restimulation, and Luminex multiplex cytokine analysis in cell culture supernatant of PBMC after restimulation with influenza viral antigens.

SECONDARY OUTCOMES:
Sleep survey - Pittsburgh Sleep Quality Index (PSQI) | 14-21 days post vaccination
  PSQI and vaccine immunogenicity (primary outcomes)
Actigraph data | 14-21 days post vaccination
  Correlation of actigraph data and vaccine immunogenicity (primary outcomes)
Chronotype survey - Munich ChronoType Questionaire (MCTQ) | 14-21 days post vaccination
  Correlation of MCTQ score with vaccine immunity

CONTACTS AND LOCATIONS:
Overall Officials: Janine Danko, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Naval Support Activity, Bethesda, Maryland, United States